CLINICAL TRIAL: NCT03914625
Title: A Phase 3 Trial Investigating Blinatumomab (NSC# 765986) in Combination With Chemotherapy in Patients With Newly Diagnosed Standard Risk or Down Syndrome B-Lymphoblastic Leukemia (B-ALL) and the Treatment of Patients With Localized B-Lymphoblastic Lymphoma (B-LLy)
Brief Title: A Study to Investigate Blinatumomab in Combination With Chemotherapy in Patients With Newly Diagnosed B-Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-02187; NCI-2019-02187 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL1731 (Other: Children's Oncology Group); AALL1731 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: B Acute Lymphoblastic Leukemia; B Lymphoblastic Lymphoma; Down Syndrome
MeSH Terms: conditions — Burkitt Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Down Syndrome | interventions — asparaginase erwinia chrysanthemi recombinant; Asparaginase; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Prednisolone; Methylprednisolone; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm A (SR-Avg control) (Active Comparator): Arm A: See detailed description.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisone; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm B (SR-Avg experimental) (Experimental): Arm B: See detailed description.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Biological: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm C (SR-High Control) (Active Comparator): Arm C: See detailed description.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Prednisone; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm D (SR-High experimental) (Experimental): Arm D See detailed description.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Biological: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Prednisone; Drug: Thioguanine; Drug: Vincristine Sulfate
- B-LLy (Experimental): See detailed description.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Prednisone; Drug: Thioguanine; Drug: Vincristine Sulfate
- DS B-ALL (Experimental): See detailed description.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Pegaspargase; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate
- NCI SR or HR DS B-ALL (Experimental): See detailed description.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Biological: Blinatumomab; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Drug: Prednisone; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Asparaginase Erwinia chrysanthemi — Given IV or IM
  Other Names: Asparaginase Erwinia chrysanthemi (Recombinant)-rywn; Asparaginase Erwinia chrysanthemi, Recombinant-rywn; Asparaginase Erwinia chrysanthemi-rywn; Crisantaspase; Crisantaspase Biobetter JZP-458; Crisantaspasum; Enrylaze; Erwinase; Erwinaze; JZP 458; JZP-458; JZP458; PF743; RC-P JZP-458; Recombinant Asparaginase erwinia chrysanthemi JZP-458; Recombinant Crisantaspase JZP-458; Recombinant Erwinia asparaginase JZP-458; Rylaze
Biological: Blinatumomab — Given IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
  Arms: Arm B (SR-Avg experimental); Arm D (SR-High experimental); NCI SR or HR DS B-ALL
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Arm A (SR-Avg control); Arm B (SR-Avg experimental); Arm C (SR-High Control); Arm D (SR-High experimental); B-LLy; DS B-ALL
Drug: Cytarabine — Given IT or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm A (SR-Avg control); Arm B (SR-Avg experimental); Arm C (SR-High Control); Arm D (SR-High experimental); B-LLy; DS B-ALL
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Leucovorin Calcium — Given PO or IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Mercaptopurine Oral Suspension — Given PO
  Other Names: 6-MP Oral Suspension; Purixan; Xaluprine
Drug: Methotrexate — Given IT or IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pegaspargase — Given IV or IM
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisolone — Given PO or IV
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
  Arms: Arm C (SR-High Control); Arm D (SR-High experimental); B-LLy; NCI SR or HR DS B-ALL
Drug: Prednisone — Given PO or IV
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Arm A (SR-Avg control); Arm C (SR-High Control); Arm D (SR-High experimental); B-LLy; NCI SR or HR DS B-ALL
Radiation: Radiation Therapy — Undergo cranial radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: DS B-ALL
Radiation: Radiation Therapy — Undergo testicular radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: DS B-ALL
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
  Arms: Arm A (SR-Avg control); Arm B (SR-Avg experimental); Arm C (SR-High Control); Arm D (SR-High experimental); B-LLy; DS B-ALL
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase III trial studies how well blinatumomab works in combination with chemotherapy in treating patients with newly diagnosed, standard risk B-lymphoblastic leukemia or B-lymphoblastic lymphoma with or without Down syndrome. Monoclonal antibodies, such as blinatumomab, may induce changes in the body's immune system and may interfere with the ability of cancer cells to grow and spread. Chemotherapy drugs, such as vincristine, dexamethasone, prednisone, prednisolone, pegaspargase, methotrexate, cytarabine, mercaptopurine, doxorubicin, cyclophosphamide, and thioguanine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Leucovorin decreases the toxic effects of methotrexate. Giving monoclonal antibody therapy with chemotherapy may kill more cancer cells. Giving blinatumomab and combination chemotherapy may work better than combination chemotherapy alone in treating patients with B-ALL. This trial also assigns patients into different chemotherapy treatment regimens based on risk (the chance of cancer returning after treatment). Treating patients with chemotherapy based on risk may help doctors decide which patients can best benefit from which chemotherapy treatment regimens.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine in a randomized manner if the addition of 2 cycles of blinatumomab to standard therapy improves disease-free survival (DFS) in patients with standard risk (SR) B-ALL and higher risk features (SR-High), and patients with standard-risk average (SR-Avg) B-ALL who are negative for minimal residual disease (MRD) by flow cytometry but have detectable or indeterminate MRD as measured by high-throughput sequencing (HTS) at end of induction (EOI).

II. To confirm that boys in the standard-risk favorable (SR-Fav) subset of B-ALL, with or without Down syndrome (DS), will maintain a 5-year DFS of greater than 93% when treated with a standard chemotherapy regimen with a treatment duration of 2 years from the start of interim maintenance I (IM1).

SECONDARY OBJECTIVES:

I. To describe the DFS for patients with SR-Avg B-ALL who are negative for MRD measured by flow cytometry and HTS at EOI when treated with standard chemotherapy with a treatment duration of 2 years from the start of IM1, regardless of sex.

II. To describe the DFS for patients with standard-risk favorable (SR-Fav) B-ALL when treated with a standard chemotherapy regimen.

III. To determine if patients with DS-High achieve a reduction of treatment-related mortality (TRM) after replacement of intensive elements of standard chemotherapy (omission of anthracyclines in induction, omission of the second month of delayed intensification [DI]) with 3 cycles of blinatumomab.

IV. To describe the DFS characterized by the replacement of intensive elements of standard chemotherapy with 3 cycles of blinatumomab in patients with DS-High B ALL.

V. To describe the DFS for patients with localized (Murphy stage I and II) B lymphoblastic lymphoma (B-LLy) receiving standard risk B-ALL therapy.

VI. To compare the change in neurocognitive functioning, as measured by the CogState Cognitive Composite, from baseline to end-of-therapy among patients with ALL ages 4- < 10 years at the time of diagnosis between children from poor families (defined as presence of household material hardship [HMH], including either food, housing or energy insecurity) and non-poor families (absence of HMH).

VII. To describe the impact of blinatumomab on caregiver burden and patient/proxy-reported symptoms among a subset of children enrolled in the HMH and neurocognitive outcome study.

VII. To evaluate available peripheral blood (PB) samples at EOI using HTS MRD and compare the results against bone marrow (BM) results.

IX. To evaluate available end of Consolidation (EOC) BM samples using HTS in patients who were Day 29 MRD positive by flow cytometry and who have submitted EOC BM flow cytometry results.

EXPLORATORY OBJECTIVES:

I. To explore adaptive and innate immune functions and host genetic factors associated with severe infectious complications in children with DS B-ALL.

II. To explore the impact of acute lymphoblastic leukemia (ALL) and its therapy on neurocognitive, functional, and quality of life outcomes in patients with DS and ALL, as measured by caregiver (parent/legal guardian) questionnaires.

III. To define the prevalence of minimal marrow disease (MMD) in B-LLy and to correlate MMD at diagnosis with outcome in patients with B-LLy.

IV. To explore the significance of and genomic landscape of Ig clonal composition in pediatric B-ALL.

V. To explore the incidence of HTS MRD ≥ 0.01% versus (vs.) HTS MRD < 0.01% in patients with multiparameter flow cytometry defined MRD < 0.01% at end of Induction and genetically characterize those with discordance defined by the 0.01% threshold.

OUTLINE: All patients are assigned to, and complete an INDUCTION treatment regimen. Patients are then assigned to a CONSOLIDATION treatment regimen. Finally, following CONSOLIDATION, patients are either assigned or randomized to 1 of 7 arms.

NON-DS SR B-ALL INDUCTION: Patients receive cytarabine intrathecally (IT) on day 1, vincristine intravenous (IV) push over 1 minute on days 1, 8, 15, and 22, dexamethasone orally (PO) or IV twice daily (BID) on days 1-28, pegaspargase IV over 1-2 hours or intramuscularly (IM) on day 4, and methotrexate IT on days 8 and 29. CNS2 patients also receive cytarabine IT twice weekly except during weeks when days 8 and 29 methotrexate is administered. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.

* After Non-DS SR B-ALL INDUCTION, SR-Fav and SR-Avg patients complete SR CONSOLIDATION, while patients with SR-High complete high-risk (HR) CONSOLIDATION.

DS B-ALL INDUCTION: Patients receive cytarabine IT on day 1, vincristine IV push over 1 minute on days 1, 8, 15, and 22, pegaspargase IV over 1-2 hours or IM on day 4, methotrexate IT on days 8 and 29, and leucovorin PO or IV every 6 hours for 2 doses on days 9 and 30. Additionally, patients under 10 years of age receive dexamethasone PO or IV BID on days 1-28, and patients 10 years of age or older receive prednisone or prednisolone PO or IV BID on days 1-28. CNS2 patients also receive cytarabine IT twice weekly except during weeks when days 8 and 29 IT methotrexate is administered. CNS3 patients also receive methotrexate IT on days 15 and 22, and leucovorin PO or IV every 6 hours for 2 doses on days 16 and 23. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.

* After DS B-ALL INDUCTION, patients without high risk features and MRD < 0.01 % complete SR CONSOLIDATION. Patients without high risk features and MRD >= 0.01%, OR with high risk features and any MRD complete HR CONSOLIDATION.

NON-DS B-LLy INDUCTION: Patients receive cytarabine IT on day 1 and twice weekly if CNS2, vincristine IV push over 1 minute on days 1, 8, 15, and 22, dexamethasone PO or IV BID on days 1-28, pegaspargase IV over 1-2 hours or IM on day 4, and methotrexate IT on days 8 and 29. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.

* After NON-DS B-LLy INDUCTION, all B-LLy patients then complete SR CONSOLIDATION.

DS B-LLY INDUCTION: Patients receive cytarabine IT on day 1, vincristine IV push over 1 minute on days 1, 8, 15, and 22, pegaspargase IV over 1-2 hours or IM on day 4, methotrexate IT on days 8 and 29, and leucovorin PO or IV every 6 hours for 2 doses on days 9 and 30. Additionally, patients under 10 years of age receive dexamethasone PO or IV BID on days 1-28, and patients 10 years of age or older receive PO or IV prednisone or methylprednisolone on days 1-28. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.

* After DS B-LLy INDUCTION, patients then complete SR CONSOLIDATION.

SR CONSOLIDATION: Patients receive vincristine IV push over 1 minute on day 1, mercaptopurine PO on days 1-28, and methotrexate IT on days 1, 8, and 15. DS patients also receive leucovorin PO or IV every 6 hours for 2 doses on days 2, 9, and 16. Treatment continues for 28 days in the absence of disease progression or unacceptable toxicity.

* After SR CONSOLIDATION, patients with MRD undetectable are assigned to ARM A, and patients with MRD detectable/indeterminate/unavailable are randomized to ARM A or B. Patients with SR-Fav and all B-LLy patients are assigned to treatments identical to that in ARM A.

HR CONSOLIDATION: Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine IV over 1-30 minutes or SC on days 1-4, 8-11, 29-32, and 36-39, vincristine IV push over 1 minute on days 15, 22, 43, and 50, mercaptopurine PO on days 1-14 and 29-42, methotrexate IT on days 1, 8, 15, and 22 , and pegaspargase IV over 1-2 hours or IM on days 15 and 43. DS patients also receive leucovorin PO or IV every 6 hours for 2 doses on days 2, 9, 16, and 23 (on days 2 and 9 only for DS CNS3 patients). Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity. Patients with continued clinical evidence of DS or testicular leukemia (from diagnosis through the end of Induction) undergo testicular radiation therapy over 12 fractions once daily (QD).

* After HR CONSOLIDATION, patients are randomized to ARM C or D. DS B-ALL patients with MRD < 1% are assigned to an arm including three blocks of blinatumomab.

ARM A:

* INTERIM MAINTENANCE I: Patients receive vincristine IV push over 1 minute on days 1, 11, 21, 31, and 41, methotrexate IV over 2-5 minutes (undiluted) or 10-15 minutes (diluted) on days 1, 11, 21, 31, and 41, and methotrexate IT on day 31. DS patients also receive leucovorin PO or IV every 6 hours for 2 doses on day 32. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* DELAYED INTENSIFICATION: Patients receive methotrexate IT on day 1 and 29, dexamethasone PO BID or IV on days 1-7 and 15-21, vincristine IV push over 1 minute on days 1, 8, and 15, doxorubicin IV push/infusion over 1-15 minutes on days 1, 8, and 15, pegaspargase IV over 1-2 hours or IM on day 4, cyclophosphamide IV over 30-60 minutes on day 29, thioguanine PO on days 29-42, and cytarabine IV over 1-30 minutes or subcutaneously (SC) on days 29-32 and 36-39. DS patients receive leucovorin PO or IV every 6 hours for 2 doses on days 2 and 30. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* INTERIM MAINTENANCE II: Patients receive vincristine IV push over 1 minute on days 1, 11, 21, 31, and 41, methotrexate IV over 2-5 minutes undiluted or 10-15 minutes diluted on days 1, 11, 21, 31, and 41, and methotrexate IT on days 1 and 31. DS patients receive leucovorin PO or IV every 6 hours for 2 doses on days 2 and 32. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* MAINTENANCE: Non-DS patients receive methotrexate IT on day 1, vincristine IV push over 1 minute on day 1, dexamethasone PO on days 1-5, mercaptopurine PO on days 1-84, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78. DS patients receive vincristine IV push over 1 minute on day 1, methotrexate IT on day 1, dexamethasone PO on days 1-5, mercaptopurine PO on days 1-84, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78, and leucovorin IV or PO on day 2 if DS. Treatment repeats every 84 days until a total duration of therapy of 2 years from start of INTERIM MAINTENANCE I is reached in the absence of disease progression or unacceptable toxicity.

ARM B:

* BLINATUMOMAB BLOCK I: Patients receive dexamethasone IV or PO on day 1, methotrexate IT on day 1, and blinatumomab IV continuously on days 1-28. DS patients also receive leucovorin IV or PO every 6 hours for 2 doses on day 2. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.
* INTERIM MAINTENANCE I: Patients receive vincristine IV push over 1 minute on days 1, 11, 21, 31, and 41, methotrexate IV over 2-5 minutes (undiluted) or 10-15 minutes (diluted) on days 1, 11, 21, 31, and 41, and methotrexate IT on day 31. DS patients also receive leucovorin PO or IV every 6 hours for 2 doses on day 32. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* BLINATUMOMAB BLOCK II: Patients receive methotrexate IT on day 1, and blinatumomab IV continuously on days 1-28. DS patients also receive leucovorin PO or IV every 6 hours for 2 doses on day 2. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.
* DELAYED INTENSIFICATION: Patients receive methotrexate IT on day 1 and 29, dexamethasone PO or IV on days 1-7 and 15-21, vincristine IV push over 1 minute on days 1, 8, and 15, doxorubicin IV push/infusion over 1-15 minutes on days 1, 8, and 15, pegaspargase IV over 1-2 hours or IM on day 4, cyclophosphamide IV over 30-60 minutes on day 29, thioguanine PO on days 29-42, and cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39. DS patients receive leucovorin PO or IV every 6 hours for 2 doses on days 2 and 30. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* INTERIM MAINTENANCE II: Patients receive vincristine IV push over 1 minute on days 1, 11, 21, 31, and 41, methotrexate IV over 2-5 minutes (undiluted) or 10-15 minutes (diluted) on days 1, 11, 21, 31, and 41, and methotrexate IT on days 1 and 31. DS patients also receive leucovorin PO or IV every 6 hours for 2 doses on days 2 and 32. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* MAINTENANCE: Non-DS patients receive methotrexate IT on day 1 (omit cycles 5-6), vincristine IV push over 1 minute on day 1, dexamethasone PO on days 1-5, mercaptopurine PO on days 1-84, and methotrexate PO on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 (omit day 1 when coinciding with IT methotrexate). DS patients receive methotrexate IT on day 1 (omit cycles 5-6), dexamethasone PO on days 1-5, mercaptopurine PO on days 1-84, and methotrexate PO on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 (omit day 1 when coinciding with IT methotrexate), for DS patients and leucovorin IV or PO every 6 hours for 2 doses on day 2 (omit on final 2 cycles). Treatment repeats every 84 days until a total duration of therapy of 2 years from start of INTERIM MAINTENANCE I is reached in the absence of disease progression or unacceptable toxicity.

ARM C:

* INTERIM MAINTENANCE I: Patients receive vincristine IV push over 1 minute on days 1, 15, 29, and 43, high dose methotrexate IV on days 1, 15, 29, and 43, mercaptopurine PO on days 1-14, 15-28, 29-42, and 43-56, methotrexate IT on day 1 and 29, and leucovorin PO or IV on days 3-4, 17-18, 31-32, and 45-46. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* DELAYED INTENSIFICATION: Patients receive methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-7 and 15-21, vincristine IV over 1 minute on days 1, 8, 15, 43, and 50, doxorubicin IV over 1-15 minutes on days 1, 8, and 15, pegaspargase IV over 1-2 hours or IM on days 4 and 43, cyclophosphamide IV over 30-60 minutes on day 29, thioguanine PO on days 29-42, and cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* INTERIM MAINTENANCE II: Patients receive vincristine IV over 1 minute on days 1, 11, 21, 31, and 41, Capizzi style methotrexate IV over 2-5 minutes (undiluted) or over 10-15 minutes (diluted) on days 1, 11, 21, 31, and 41, methotrexate IT on days 1 and 31, and pegaspargase IV over 1-2 hours or IM on days 2 and 22. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* MAINTENANCE: Patients receive vincristine IV over 1 minute on day 1, prednisone or prednisolone or methylprednisolone PO or IV on days 1-5, mercaptopurine PO on days 1-84, methotrexate IT on days 1 and 29 of cycles 1-2 and on day 1 of subsequent cycles, methotrexate PO on days 8, 15, 22, 29 (for cycle 3 and later only), 36, 43, 50, 57, 64, 71, and 78. Treatment repeats every 84 days until a total duration of therapy of 2 years from start of interim maintenance I is reached in the absence of disease progression or unacceptable toxicity.

ARM D:

* BLINATUMOMAB BLOCK I: Patients receive dexamethasone PO or IV on day 1, methotrexate IT on day 1, and blinatumomab IV continuously on days 1-28. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.
* INTERIM MAINTENANCE I: Patients receive vincristine IV over 1 minute on days 1, 15, 29, and 43, high dose methotrexate IV on days 1, 15, 29, and 43, mercaptopurine PO on days 1-14, 15-28, 29-42, and 43-56, methotrexate IT on days 1 and 29, and leucovorin PO or IV on days 3-4, 17-18, 31-32, and 45-46. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* BLINATUMOMAB BLOCK II: Patients receive blinatumomab IV on days 1-28 and methotrexate IT on day 1. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.
* DELAYED INTENSIFICATION: Patients receive methotrexate IT on day 1, dexamethasone PO or IV on days 1-7 and 15-21, vincristine IV over 1 minute on days 1, 8, 15, 43, and 50, doxorubicin IV over 1-15 minutes on days 1, 8, and 15, pegaspargase IV over 1-2 hours or IM on days 4 and 43, cyclophosphamide IV over 30-60 minutes on day 29, thioguanine PO on days 29-42, and cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* INTERIM MAINTENANCE II: Patients receive vincristine IV over 1 minute on days 1, 11, 21, 31, and 41, Capizzi style methotrexate IV over 2-5 minutes (undiluted) or over 10-15 minutes (diluted) on days 1, 11, 21, 31, and 41, methotrexate IT on days 1 and 31, and pegaspargase IV over 1-2 hours or IM on days 2 and 22. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* MAINTENANCE: Patients receive methotrexate IT on day 1, vincristine IV over 1 minute on day 1, prednisone, prednisolone or methylprednisolone PO or IV on days 1-5, mercaptopurine PO on days 1-84, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78. Treatment repeats every 84 days until a total duration of therapy of 2 years from start of interim maintenance I is reached in the absence of disease progression or unacceptable toxicity.

DS-HIGH B-ALL:

* BLINATUMOMAB BLOCK I: Patients receive dexamethasone PO or IV on day 1, blinatumomab IV continuously on days 1-28, methotrexate IT on day 1 (or on day 56 of Consolidation), and leucovorin PO or IV every 6 hours for 2 doses on day 2. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.
* INTERIM MAINTENANCE: Patients receive vincristine IV push over 1 minute on days 1, 15, 29, and 43, intermediate dose methotrexate IV over 24 hours on days 1, 15, 29, and 43, mercaptopurine PO on days 1-14, 15-28, 29-42, and 43-46, methotrexate IT on days 1 and 29, and leucovorin PO or IV every 6 hours for 2 doses on days 2-4, 16-18, 30-32, and 44-46. Treatment continues for 63 days in the absence of disease progression or unacceptable toxicity.
* BLINATUMOMAB BLOCK II: Patients receive blinatumomab IV on days 1-28, methotrexate IT on day 1, and leucovorin PO or IV every 6 hours for 2 doses on day 2. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.
* DELAYED INTENSIFICATION: Patients receive vincristine IV over 1 minute on days 1, 8, and 15, doxorubicin IV over 1-15 minutes on days 1, 8, and 15, dexamethasone PO or IV on days 1-7 and 15-21, methotrexate IT on day 1, leucovorin PO or IV every 6 hours for 2 doses on day 2, and pegaspargase IV over 1-2 hours or IM on day 4. Treatment continues for 28 days in the absence of disease progression or unacceptable toxicity.
* BLINATUMOMAB BLOCK III: Patients receive blinatumomab IV on days 1-28, methotrexate IT on day 1, and leucovorin PO or IV every 6 hours for 2 doses on day 2. Treatment continues for 35 days in the absence of disease progression or unacceptable toxicity.
* MAINTENANCE: Patients receive vincristine IV push over 1 minute on day 1, prednisone, prednisolone or methylprednisolone PO or IV BID on days 1-5, mercaptopurine PO on days 1-84, methotrexate IT on day 1, methotrexate PO on days 8, 15, 22, 29 (omit day 29 for first 3 cycles for patients who do not receive cranial radiotherapy), 36, 43, 50, 57, 64, 71, and 78, and leucovorin PO on days 2 and 30 (day 30 dose is for cycles 1-3 and for patients who do not receive cranial radiotherapy). CNS3 patients receive cranial radiotherapy during first 4 weeks of cycle 1. Treatment repeats every 84 days until a total duration of therapy of 2 years from start of interim maintenance I is reached in the absence of disease progression or unacceptable toxicity.

All B-LLy patients:

* INTERIM MAINTENANCE I: Patients receive vincristine IV push over 1 minute on days 1, 11, 21, 31, and 41, methotrexate IV over 2-5 minutes (undiluted) or 10-15 (diluted) on days 1, 11, 21, 31, and 41, and methotrexate IT on day 31. DS patients also receive leucovorin PO or IV every 6 hours for 2 doses on day 32. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* DELAYED INTENSIFICATION: Patients receive vincristine IV push over 1 minute on days 1, 8 and 15, doxorubicin IV over 1-15 minutes on days 1, 8, and 15, dexamethasone PO or IV on days 1-7 and 15-21, methotrexate IT on days 1 and 29, pegaspargase IV over 1-2 hours or IM on day 4, cyclophosphamide IV over 30-60 minutes on day 29, thioguanine PO on days 29-42, and cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39. DS patients additionally receive leucovorin PO or IV every 6 hours for 2 doses on days 2 and 30. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* INTERIM MAINTENANCE II: Patients receive vincristine IV push over 1 minute on days 1, 11, 21, 31, and 41, methotrexate IV over 2-5 minutes (undiluted) or 10-15 minutes (diluted) on days 1, 11, 21, 31, and 41, and methotrexate IT on days 1 and 31. DS patients also receive leucovorin PO or IV every 6 hours for 2 doses on days 2 and 32. Treatment continues for 56 days in the absence of disease progression or unacceptable toxicity.
* MAINTENANCE: Patients receive vincristine IV push over 1 minute on day 1, dexamethasone PO on days 1-5, mercaptopurine PO on days 1-84, methotrexate IT on day 1, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78. DS patients also receive leucovorin PO or IV every 6 hours for 2 doses on day 2. Treatment repeats every 84 days until a total duration of therapy of 2 years from start of interim maintenance I is reached in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 weeks until complete blood count(CBC)/differential/platelet count recovery, then every 3 months for the first 2 years, then every 4-6 months for the 3rd year, and every 6-12 months for the 4th and 5th years.

ELIGIBILITY:
Inclusion Criteria:

* All B-ALL patients must be enrolled on APEC14B1 and consented to Eligibility Screening (Part A) prior to treatment and enrollment on AALL1731. APEC 14B1 is not a requirement for B-LLy patients. B-LLy patients may directly enroll on AALL1731.
* Age at diagnosis:

  * Patients must be >= 365 days and < 10 years of age (B-ALL patients without DS).
  * Patients must be >= 365 days and =< 31 years of age (B-ALL patients with DS).
  * Patients must be >= 365 days and =< 31 years of age (B-LLy patients with or without DS).
* B-ALL patients without DS must have an initial white blood cell count < 50,000/uL (performed within 7 days prior to enrollment).
* B-ALL patients with DS are eligible regardless of the presenting white blood cell count (WBC) (performed within 7 days prior to enrollment).
* Patient has newly diagnosed B-cell ALL, with or without Down syndrome: > 25% blasts on a bone marrow (BM) aspirate;

  * OR if a BM aspirate is not obtained or is not diagnostic of B-ALL, the diagnosis can be established by a pathologic diagnosis of B-ALL on a BM biopsy;
  * OR a complete blood count (CBC) documenting the presence of at least 1,000/uL circulating leukemic cells;
  * OR patient has newly diagnosed B-cell LLy Murphy stages I or II, with or without Down syndrome.
  * Note: For B-LLy patients with tissue available for flow cytometry, the criterion for diagnosis should be analogous to B-ALL. For tissue processed by other means (i.e., paraffin blocks), the methodology and criteria for immunophenotypic analysis to establish the diagnosis of B-LLy defined by the submitting institution will be accepted (diagnostic biopsy for B-LLy must be performed within 14 days prior to enrollment).
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* Patient must not have secondary ALL that developed after treatment of a prior malignancy with cytotoxic chemotherapy. Note: patients with Down syndrome with a prior history of transient myeloproliferative disease (TMD) are not considered to have had a prior malignancy. They would therefore be eligible whether or not the TMD was treated with cytarabine.
* With the exception of steroid pretreatment or the administration of intrathecal cytarabine, patients must not have received any prior cytotoxic chemotherapy for either the current diagnosis of B ALL or B LLy or for any cancer diagnosed prior to initiation of protocol therapy on AALL1731.
* For patients receiving steroid pretreatment, the following additional exclusion criteria apply:

  * Non-DS B-ALL patients must not have received steroids for more than 24 hours in the 2 weeks prior to diagnosis without a CBC obtained within 3 days prior to initiation of the steroids.
  * DS and non-DS B-LLy patients must not have received > 48 hours of oral or IV steroids within 4 weeks of diagnosis.
* Patients who have received > 72 hours of hydroxyurea within 1 week (7 days) prior to the start of systemic protocol therapy.
* B-ALL patients who do not have sufficient diagnostic bone marrow submitted for APEC14B1 diagnostic testing and who do not have a peripheral blood sample submitted containing > 1,000/uL circulating leukemia cells.
* Patient must not have acute undifferentiated leukemia (AUL).
* Non-DS B-ALL patients with central nervous system [CNS]3 leukemia (CNS status must be known prior to enrollment).

  * Note: DS patients with CNS3 disease are eligible but will be assigned to the DS-High B-ALL arm. CNS status must be determined based on a sample obtained prior to administration of any systemic or intrathecal chemotherapy, except for steroid pretreatment.
* Non-DS B-ALL patients with testicular leukemia. (Note: DS patients with testicular disease are eligible but will be assigned to the DS-High B-ALL arm).
* For LLy patients, the following additional exclusion criteria apply:

  * T-Lymphoblastic Lymphoma.
  * Morphologically unclassifiable lymphoma.
  * Absence of both B-cell and T-cell phenotype markers in a case submitted as lymphoblastic lymphoma.
  * CNS positive disease or testicular involvement.
  * M2 (5% - 25% blasts) or M3 (> 25% blasts) marrow.
* Patients with known Charcot-Marie-Tooth disease.
* Patients with known MYC translocation associated with mature (Burkitt) B-cell ALL, regardless of blast immunophenotype.
* Patients requiring radiation at diagnosis.
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential.
* Lactating females who plan to breastfeed their infants.
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation.

Ages: 365 Days to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6720 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) in randomization eligible patients with higher risk features (SR-High) or standard risk average (SR-Avg) B-ALL patients based on randomization with addition of blinatumomab | 5.3 years
  Will be assessed in SR-High patients and SR-Avg B-ALL patients who are negative for MRD by flow cytometry but have detectable or indeterminate MRD as measured by high throughput sequencing (HTS) at end of induction (EOI), and patients with double trisomy of chromosomes 4 and 10 (DT) with MRD (flow) 0.01% - < 0.1%. DFS is calculated as the time from randomization at the end of consolidation to first event (relapse, second malignancy, remission death) or censored at date of last contact. Five year DFS estimates will be calculated from the point of randomization for both groups. Two-sided 95% confidence intervals will be calculated.
DFS in boys in the SR-favorable subset of SR B-ALL with or without Down syndrome (DS) | 5.1 years
  DFS is calculated as the time from end of induction to first event (relapse, second malignancy, remission death) or censored at date of last contact. A five year DFS estimate and two-sided 80% confidence interval will be calculated.

SECONDARY OUTCOMES:
DFS for patients with SR-Avg B-ALL who are negative for MRD measured by flow cytometry and HTS at EOI when treated with standard chemotherapy with a treatment duration of 2 years from the start of interim maintenance (IM)1, regardless of sex | 5.1 years
  DFS is calculated as the time from end of induction to first event (relapse, second malignancy, remission death) or censored at date of last contact. A five year DFS estimate and a two-sided 95% confidence interval will be calculated.
DFS for patients with standard-risk favorable (SR-Fav) B-ALL when treated with a standard chemotherapy regimen | 5.1 years
  DFS is calculated as the time from end of induction to first event (relapse, second malignancy, remission death) or censored at date of last contact. A five year DFS estimate and a two-sided 95% confidence interval will be calculated.
Treatment-related mortality in Down syndrome high risk (DS-high) patients after replacement of intensive elements of standard chemotherapy (omission of anthracyclines in induction, omission of the second month of DI) with 3 cycles of blinatumomab | 2.3 years
  Percent of DS-high patients with treatment related mortalities will be reported with 95% confidence interval.
DFS of DS-High B-ALL patients when intensive elements of chemotherapy are replaced with 3 cycles of blinatumomab | 5.3 years
  DFS is calculated as the time from the end of consolidation to first event (relapse, second malignancy, remission death) or censored at date of last contact. A five year DFS estimate and a two-sided 80% confidence interval will be calculated.
DFS of patients with localized B-lymphoblastic lymphoma (B-LLy) receiving standard risk acute lymphoblastic leukemia therapy | 5 years
  DFS is calculated as the time from study enrollment to first event (disease progression, relapse, second malignancy, remission death) or censored at date of last contact. A five year DFS estimate and a two-sided 95% confidence interval will be calculated.
Change in neurocognitive functioning from baseline to end-of-therapy between children from poor (defined as presence of household material hardship [HMH], including either food, housing or energy insecurity) and non-poor families (absence of HMH) | 3.3 years
  Neurocognitive functioning will be measured by the CogState Cognitive Composite at end of induction therapy and at follow-up one year off-therapy among patients with ALL ages 4-< 10 years at the time of diagnosis. Mean and 95% confidence interval for change scores will be reported by HMH group.
Caregiver burden as measured by the Mean Total score from the Care of My Child with Cancer questionnaire among a subset of children enrolled in the HMH and neurocognitive outcome study | 1 year
  The Mean Total score from the Care of My Child with Cancer questionnaire from end of Maintenance Cycle 1. Mean scores and 95% confidence intervals will be reported by randomization group.
Caregiver burden as measured by the At-Work Productivity Loss summary score from the Caregiver Work Limitations questionnaire among a subset of children enrolled in the HMH and neurocognitive outcome study | 1 year
  The Mean Total score from the Care of My Child with Cancer questionnaire from end of Maintenance Cycle 1. Mean scores and 95% confidence intervals will be reported by randomization group.
Peripheral blood (PB) samples using HTS MRD vs. bone marrow (BM) results at EOI | 1 year
  Will use the Kendall's Tau-b rank correlation coefficient accounting for the left censoring inherent to sensitivity of the method. A high positive value would be strong evidence that the PB retains the relative information contained in the BM readings. An estimate and two-sided 95% Confidence interval will be calculated using banked SR-Average and SR-High samples at EOI.
BM using HTS MRD vs. BM by flow cytometry at EOC in patients who were Day 29 MRD positive by flow cytometry | 1 year
  Will use the Kendall's Tau-b rank correlation coefficient accounting for the left censoring inherent to sensitivity of the methods30. A high positive value would be strong evidence that HTS of IgH loci determined-MRD from the BM at EOC retains the relative information contained in the flow-cytometry-determined readings. An estimate and 95% Confidence interval will be calculated using pairs of banked samples at EOC.

OTHER OUTCOMES:
To explore adaptive and innate immune functions and host genetic factors associated with severe infectious complications in children with DS B-ALL | 5 years
  FlowSom high resolution clustering approach to identify cellular subsets and/or activation states (endophenotypes) that distinguish cases from controls. Perform secondary analysis using the "diffCyt" framework to identify those cell clusters that differ significantly between groups.
Neurocognitive, functional, and quality of life outcomes in patients with DS and ALL | 5 years
  Measured by caregiver (parent/legal guardian) using questionnaires that rate executive function, behavior, adaptive skills, and quality of life.
Prevalence of minimal marrow disease (MMD) in B-LLy | 5 years
  Correlate MMD at diagnosis with outcome in patients with B-LLy.
Genetic landscape of B-ALL lacking a clonal Ig sequence | 5 years
  Will be measured by performing targeted sequencing (hemoglobin [heme] deoxyribonucleic acid [DNA] mutation and ribonucleic acid [RNA] fusion panels) on samples from all identified patients without a clonal Ig sequence with banked material and compare to matched subjects with clonal Ig sequences. Will determine associations between having or lacking a clonal Ig sequence and discrete mutations/fusions using Fisher's exact test. Will also be assessed with a 1-sided alpha of 0.05, a log-rank test.
Association between flow cytometry | At the end of induction
  Will be determined by MRD and HTS of IgH loci from the BM in NCI SR B-ALL patients who are MRD positive by flow cytometry. Will use the Kendall's Tau-b rank correlation coefficient accounting for the left censoring inherent to sensitivity of the methods. A high positive value would be strong evidence that the PB retains the relative information contained in the BM readings. An estimate and two-sided 95% Confidence interval will be calculated using banked SR-Average and SR-High samples.

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Gupta, Principal Investigator — Children's Oncology Group
Locations (228):
- United States (201):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Palms West Radiation Therapy, Loxahatchee Groves, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Vannie Cook Children's Clinic, McAllen, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (2):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - University Pediatric Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Gupta S, Rau RE, Kairalla JA, Rabin KR, Wang C, Angiolillo AL, Alexander S, Carroll AJ, Conway S, Gore L, Kirsch I, Kubaney HR, Li AM, McNeer JL, Militano O, Miller TP, Moyer Y, O'Brien MM, Okada M, Reshmi SC, Shago M, Wagner E, Winick N, Wood BL, Haworth-Wright T, Zaman F, Zugmaier G, Zupanec S, Devidas M, Hunger SP, Teachey DT, Raetz EA, Loh ML. Blinatumomab in Standard-Risk B-Cell Acute Lymphoblastic Leukemia in Children. N Engl J Med. 2025 Feb 27;392(9):875-891. doi: 10.1056/NEJMoa2411680. Epub 2024 Dec 7. PMID 39651791
- [Derived] Sora F, Annunziata M, Laurenti L, Giammarco S, Chiusolo P, Innocenti I, Autore F, Metafuni E, Galli E, Bacigalupo A, Ferrara F, Sica S. Blinatumomab as a successful and safe therapy in Down syndrome patients with relapsed/refractory b-precursor acute lymphoblastic leukaemia: Case reports and literature review. Pediatr Blood Cancer. 2021 Jul;68(7):e29044. doi: 10.1002/pbc.29044. Epub 2021 Apr 12. No abstract available. PMID 33844429

DOCUMENTS (3):
  • Informed Consent Form: Consent B-LLy (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03914625/ICF_000.pdf
  • Informed Consent Form: Consent B-ALL (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03914625/ICF_001.pdf
  • Informed Consent Form: Consent DS-High Post Induction (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03914625/ICF_002.pdf